CLINICAL TRIAL: NCT04912492
Title: Promoting Prosocial Bystander Behavior in Intoxicated Men: Evaluation of RealConsent2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: University of Nebraska Lincoln (Other)
Responsible Party: Principal Investigator, Laura F Salazar, Multiple Principal Investigator, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AA027517 (NIH)
Record Dates: First submitted 2021-02-05; First posted 2021-06-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Intoxication; Sexual Violence; Helping Behavior
MeSH Terms: conditions — Alcoholic Intoxication; Helping Behavior | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- RealConsent 1.0 with Alcohol (Active Comparator): Men assigned to complete a web-based multi-media sexual violence and bystander intervention prevention program. Men assigned to alcohol intoxication arm (target breath alcohol concentration (BrAC=.08).
  Interventions: Behavioral: RealConsent1.0; Behavioral: Alcohol intoxication
- RealConsent 1.0 with Placebo (Active Comparator): Men assigned to complete a web-based multi-media sexual violence and bystander intervention prevention program. Men assigned to a no-alcohol placebo control arm.
  Interventions: Behavioral: RealConsent1.0; Behavioral: No-Alcohol Placebo
- RealConsent2.0 with Alcohol (Experimental): Men assigned to complete a revised web-based multi-media sexual violence and bystander intervention prevention program. Men assigned to alcohol intoxication arm (target BrAC=.08).
  Interventions: Behavioral: RealConsent2.0; Behavioral: Alcohol intoxication
- RealConsent2.0 with Placebo (Experimental): Men assigned to complete a revised web-based multi-media sexual violence and bystander intervention prevention program. Men assigned to a no-alcohol placebo control arm.
  Interventions: Behavioral: RealConsent2.0; Behavioral: No-Alcohol Placebo
- Stress Management with Alcohol (Active Comparator): Men assigned to complete a web-based stress management program. Men assigned to alcohol intoxication arm (target BrAC=.08).
  Interventions: Behavioral: Stress Management; Behavioral: Alcohol intoxication
- Stress Management with Placebo (Active Comparator): Men assigned to complete a web-based stress management program. Men assigned to a no-alcohol placebo control arm.
  Interventions: Behavioral: Stress Management; Behavioral: No-Alcohol Placebo

INTERVENTIONS:
Behavioral: RealConsent1.0 — A web-based multi-media sexual violence prevention program that enhances knowledge and skills for effective consent for sex and for prosocial bystander behaviors.
  Arms: RealConsent 1.0 with Alcohol; RealConsent 1.0 with Placebo
Behavioral: RealConsent2.0 — A revised and updated web-based multi-media sexual violence prevention program that enhances knowledge and skills for effective consent for sex and for prosocial bystander behaviors, but also integrates new program segments into RealConsent 1.0 specific to how alcohol use can inhibit SV intervention at multiple steps of the decision-making process.
  Arms: RealConsent2.0 with Alcohol; RealConsent2.0 with Placebo
Behavioral: Stress Management — A web-based multimedia program designed to help individuals recognize the symptoms and sources of stress and provide them with a wide variety of powerful tools for managing stress.
  Arms: Stress Management with Alcohol; Stress Management with Placebo
Behavioral: Alcohol intoxication — Men assigned to moderate alcohol dose condition (target BrAC .08%) with NIAAA approved alcohol administration procedures
  Arms: RealConsent 1.0 with Alcohol; RealConsent2.0 with Alcohol; Stress Management with Alcohol
Behavioral: No-Alcohol Placebo — Men assigned to an no-alcohol placebo control condition.
  Arms: RealConsent 1.0 with Placebo; RealConsent2.0 with Placebo; Stress Management with Placebo

SUMMARY:
Sexual violence (SV) is a significant public health problem particularly among 18-24 year old populations. A major risk factor for SV is alcohol use, which via its negative impact on cognitive abilities and decision-making acts as a barrier to intervening in situations at-risk for a SV. This study has two main goals: (1) to determine the effects of proximal alcohol use on young (age 21 to 25) men's prosocial bystander behavior in situations considered at-risk for SV, and (2) to determine the efficacy of an evidence-based, web-based program called RealConsent, which has been augmented to include alcohol-specific content within the context of bystander SV ("RealConsent2.0"), on men's prosocial bystander behavior. The primary study endpoint is prosocial bystander behavior and will be assessed via two modes: (1) a virtual reality (VR) environment ("B-SAVE") and (2) a validated self-report measure of bystander behavior that has been modified to include assessment of proximal alcohol use and presence of alcohol within the context.

ELIGIBILITY:
Inclusion Criteria:

* identify as a man or transgender man, age (21-25)
* consume weight-based amount of alcohol at least three times during the past year

Exclusion Criteria:

* weight over 250 pounds
* current treatment-seeking for an alcohol use disorder
* any medical or psychiatric condition, as well as current use of a medication, that would contraindicate alcohol administration.
* in a relationship over 6 months
* married/living together
* Neurological Disorder: diagnosis of a neurological disorder
* Psychiatric Disorder: past or current diagnosis of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, or any other psychotic disorder
* Treatment for Alcohol or Drug Use: currently being treated for alcohol, or drug problems; currently interested in seeking treatment for drinking or drug use
* Physical disability: anh physical disability that would prevent an individual from participating in the virtual reality task (self-report and determined)
* Significant Hearing Problems: significant hearing problems that would prevent an individual from hearing and responding to the virtual reality task (self-reported and determined)
* Cardiac Pacemaker
* Asthma: emergency room visit related to asthma in the past year; use of inhaler more frequently when drinking alcohol; use of oral steroid treatments for asthma in the past year;
* Legal: any legal restrictions against drinking (e.g., as a condition of probation or parole)
* Alcohol Abstinence: individuals who consume alcohol monthly or less; individuals who have consumed the amount of alcohol they would be expected to drink during the lab session (determined by their weight) less than 3 times in the last year
* Head Injury: any past serious head injuries (as indicated by HELPS Brain Injury Screening Tool)
* Acute Psychiatric Symptomatology: elevated psychological distress as indicated by a score greater than 65 on the Brief Symptom Inventory

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must identify as a man or transgender man
Enrollment: 667 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Bystander behavior | One-month post-intervention
  Bystander behavior will be assessed by a virtual reality (VR) environment titled, Bystanders in Sexual Assault Virtual Environments (B-SAVE). Participants experience a virtual "house party" and are exposed to 5 situations in which they can either intervene or not. Participants are prompted at two points (with a flashing microphone icon) to verbalize their response in that situation - thus providing 10 opportunities to intervene in sexual risk situations. Verbal responses to each situation are recorded and coded to assess for bystander behavior.
Self-Reported Bystander Behavior | Change from Baseline at 6-months
  The 44-item Bystander Behavior Scale involves a description of a scenario in which participants are asked if they were exposed to the scenario, did they engage in the behavior (yes/no), if they had been drinking alcohol (yes/no) and if alcohol was present (yes/ no). Response options range from 0 (no) to 1 (yes) for each of the items. A total score for bystander behavior is calculated ranging from 0 (minimum) to 30 (maximum), with higher scores indicating greater bystander behavior in the last three-months. alcohol (yes/no) and if alcohol was present (yes/ no).
Self-Reported Bystander Behavior | Change from Baseline at 12-months
  The 44-item Bystander Behavior Scale involves a description of a scenario in which participants are asked if they were exposed to the scenario, did they engage in the behavior (yes/no), if they had been drinking alcohol (yes/no) and if alcohol was present (yes/ no). Response options range from 0 (no) to 1 (yes) for each of the items. A total score for bystander behavior is calculated ranging from 0 (minimum) to 30 (maximum), with higher scores indicating greater bystander behavior in the last three-months. alcohol (yes/no) and if alcohol was present (yes/ no).

SECONDARY OUTCOMES:
Barriers to Sexual Assault Bystander Intervention | Change from Baseline at 6-months
  The 16-item Barriers to Sexual Assault Bystander Intervention Scale assess barriers to intervention. Mean scores range from 1 (minimum) to 7 (maximum), with higher scores indicate more barriers to intervention.
Barriers to Sexual Assault Bystander Intervention | Change from Baseline at 12-months
  The 16-item Barriers to Sexual Assault Bystander Intervention Scale assess barriers to intervention. Mean scores range from 1 (minimum) to 7 (maximum), with higher scores indicate more barriers to intervention.
Outcome Expectancies for Intervening | Change from Baseline at 6-months
  The 17-item Outcome Expectancies for Intervening Scale assess outcome expectancies for intervening. Mean scores ranging from 1 (minimum) to 7 (maximum). Higher scores indicate greater positive expectancies for intervening.
Outcome Expectancies for Intervening | Change from Baseline at 12-months
  The 17-item Outcome Expectancies for Intervening Scale assess outcome expectancies for intervening. Mean scores ranging from 1 (minimum) to 7 (maximum). Higher scores indicate greater positive expectancies for intervening.
Bystander Efficacy Scale | Change from Baseline at 6-months
  14-item Bystander Efficacy Scale assess bystander confidence to intervene, with response options ranging from 0 % (minimum) to 100% (maximum). A score is created by subtracting the mean of these 14 items from 100 to create a scale of perceived efficacy. Higher scores indicate greater bystander efficacy.
Bystander Efficacy Scale | Change from Baseline at 12-months
  14-item Bystander Efficacy Scale assess bystander confidence to intervene, with response options ranging from 0 % (minimum) to 100% (maximum). A score is created by subtracting the mean of these 14 items from 100 to create a scale of perceived efficacy. Higher scores indicate greater bystander efficacy.
Bystander Attitude Scale | Change from Baseline at 6-months
  The 12-item Bystander Attitudes Scale assesses bystander intentions. Response options ranging from 1 (minimum) to 5 (maximum), with greater mean scores indicate higher intentions of intervening.
Bystander Attitude Scale | Change from Baseline at 12-months
  The 12-item Bystander Attitudes Scale assesses bystander intentions. Response options ranging from 1 (minimum) to 5 (maximum), with greater mean scores indicate higher intentions of intervening.
Sexual Violence Perpetration | Change from Baseline at 6-months
  The 35 items Sexual Experience Survey will be used to assess sexual violence perpetration. Participants indicate the number of times that they did each act ranging from 0 (never) to 3 (3 or more times), with total scores ranging from 0 to 105 with greater scores indicating more perpetration. The mutually exclusive scoring system will be used. The goal is to count people only once according to the most severe act perpetrated.
Sexual Violence Perpetration | Change from Baseline at 12-months
  The 35 items Sexual Experience Survey will be used to assess sexual violence perpetration. Participants indicate the number of times that they did each act ranging from 0 (never) to 3 (3 or more times), with total scores ranging from 0 to 105 with greater scores indicating more perpetration. The mutually exclusive scoring system will be used. The goal is to count people only once according to the most severe act perpetrated.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Salazar, Ph.D., Principal Investigator — Georgia State University
Locations (2):
- United States (2):
  - Georgia State University, Atlanta, Georgia
  - University of Nebraska-Lincoln, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
After the grant period, access to the data will be provided through the Inter- University Consortium for Political and Social Research (ICPSR). Users will be required to agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data source and funders. One year after the study is completed, all data will be compiled and organized into a single repository at ICPSR. Data will be made publicly available through ICPSR's website.
Time Frame: One year after the study is completed, all data will be compiled and organized into a single repository at ICPSR.
Access Criteria: Users will be required to agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgment of the data source and funders.

REFERENCES:
- [Derived] Salazar LF, Parrott DJ, DiLillo D, Gervais S, Schipani-McLaughlin AM, Leone R, Swartout K, Simpson L, Moore R, Wilson T, Flowers N, Church H, Baildon A. Study protocol for a randomized controlled trial of RealConsent2.0: a web-based intervention to promote prosocial alcohol-involved bystander behavior in young men. Trials. 2023 Dec 12;24(1):804. doi: 10.1186/s13063-023-07797-w. PMID 38087306